CLINICAL TRIAL: NCT03567434
Title: Randomized, Double-Blind, Placebo-Based Study to Determine Effect of Evening Alcohol on Sympathetic Neural Activity and Baroreflex Function in Binge Drinkers
Brief Title: Alcohol and Neural Cardiovascular Control in Binge Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: University of Chicago (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: JC080420-FC; 1R01AA024892-01A1 (NIH)
Record Dates: First submitted 2018-05-24; First posted 2018-06-25 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Binge Drinking
MeSH Terms: conditions — Binge Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid Control (Placebo Comparator): Participants first received a fluid control drink (i.e., juice) of the same volume of fluid as the alcohol condition. After at least a one-month washout period, they then received the alcohol condition.
  Interventions: Other: Alcohol vs. Placebo
- Alcohol (Experimental): Participants first received the alcohol condition with 95% ethanol and fruit juice (1:3 ratio). After at least a one-month washout period, they then received the fluid control condition with a volume fluid match.
  Interventions: Other: Alcohol vs. Placebo

INTERVENTIONS:
Other: Alcohol vs. Placebo — Using a randomized, cross-over design, all subjects will consume evening alcohol (and a fluid-control placebo) in a dose that mimics binge drinking.
  Other Names: Ethanol

SUMMARY:
This study evaluates the impact of evening alcohol consumption on sympathetic activity and baroreflex function in binge drinkers. Our central hypothesis is that evening binge alcohol consumption will lead to sympathetic overactivity and blunted baroreflex function.

DETAILED DESCRIPTION:
This study will recruit male and female binge drinkers who will participate in a randomized, cross-over, double-blind, placebo-based study to examine the impact of an evening of alcohol vs. placebo/fluid-control on autonomic and cardiovascular control at night and the subsequent morning. The study will utilize established techniques for assessing sleep (polysomnography) and autonomic/cardiovascular control (microneurography, beat-to-beat finger plethysmography, electrocardiogram, etc.). All subjects will undergo a familiarization night in the sleep laboratory prior to their first randomized test session with either alcohol or placebo/fluid-control. Both men and women will be tested to address a secondary aim of determining the impact of sex (male vs. female) and ovarian cycle (early follicular vs. midluteal phase) on sympathetic neural responsiveness to evening alcohol in binge drinkers. Finally, as a tertiary/exploratory aim, participants that have a respiratory disturbance index of ≥5 episodes per hour during the alcohol treatment will be asked to consider one additional overnight session where they will be randomly assigned to either continuous positive airway pressure (CPAP) or sham-CPAP for one additional night of evening alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 21 - 40 years
* Binge drinkers as defined by a pattern of consuming ≥4 drinks if female (≥5 drinks if males) in ≤ 2 hours on more than one occasion within the past 6 months, and at least once in the past 30 days. The National Institute of Alcohol Abuse and Alcoholism (NIAAA) definition of a "drink" will be used.
* Women must be eumenorrheic and premenopausal with regular and consistent menstrual cycles (i.e., ~25-30 days ovarian/uterine cycles that include 2-7 days of menstruation)
* Willingness to abstain from exercise and caffeine at least 12 hours prior to any autonomic and cardiovascular testing, and abstain from alcohol 24 hours prior to any autonomic and cardiovascular testing (unless experimentally administered).

Exclusion Criteria:

* Body mass index ≥ 35 kg/m2
* Smokers
* A physician diagnosis of diabetes
* Pregnancy
* Taking any cardiovascular medications
* Severe obstructive sleep apnea as determined by an apnea-hypopnea index of ≥ 30 episodes per hour
* Moderate-to-severe Alcohol Use Disorder (AUD) as determined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-V)
* Individuals suspected to have mutant alcohol dehydrogenase 2 (ALDH2) isoenzyme as determined using a validated flushing questionnaire
* Women using hormonal contraceptives (i.e., oral, intrauterine, etc.) in the prior 6 months

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Carter, Principal Investigator — Baylor University
Locations (1):
- Montana State University, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No
The scientific field of neural cardiovascular control in humans does not, at present, have a common data repository that would be applicable to this project. However, all data will be stored on secure University server in a de-identified manner, and investigators will make raw data available to individuals, groups, and organizations upon request and when appropriate.

REFERENCES:
- [Derived] Bigalke JA, Greenlund IM, Solis-Montenegro TX, Durocher JJ, Joyner MJ, Carter JR. Binge Alcohol Consumption Elevates Sympathetic Transduction to Blood Pressure: A Randomized Controlled Trial. Hypertension. 2024 Oct;81(10):2140-2151. doi: 10.1161/HYPERTENSIONAHA.124.23416. Epub 2024 Aug 9. PMID 39119705
- [Derived] Greenlund IM, Bigalke JA, Tikkanen AL, Durocher JJ, Smoot CA, Carter JR. Evening binge alcohol disrupts cardiovagal tone and baroreflex function during polysomnographic sleep. Sleep. 2021 Nov 12;44(11):zsab130. doi: 10.1093/sleep/zsab130. PMID 34015116

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by word-of-mouth and advertisements. 169 participants were screened for eligibility.
Pre-assignment Details: 38/169 participants were randomized. Of the 131 that were not randomized 100 did not meet inclusion criteria or did not consent and 31 were lost to follow-up/drop out.
Groups:
- Fluid Control, Then Alcohol: Participants first received a fluid control drink (i.e., juice) of the same volume of fluid as the alcohol condition. After at least a one-month washout period, they then received the alcohol condition.
  Alcohol vs. Placebo: Using a randomized, cross-over design, all subjects will consume evening alcohol (and a fluid-control placebo) in a dose that mimics binge drinking.
- Alcohol, Then Fluid Control: Participants first received the alcohol condition with 95% ethanol and fruit juice (1:3 ratio). After at least a one-month washout period, they then received the fluid control condition with a volume fluid match.
  Alcohol vs. Placebo: Using a randomized, cross-over design, all subjects will consume evening alcohol (and a fluid-control placebo) in a dose that mimics binge drinking.
Period: Overall Study
Arm/Group | Fluid Control, Then Alcohol | Alcohol, Then Fluid Control
Started | 16 | 22
Completed Test 1 | 16 | 22
Completed Test 2 | 15 | 19
Completed | 15 | 19
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluid Control, Then Alcohol | Alcohol, Then Fluid Control | Total
Number analyzed (Participants) | 16 | 22 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 22 | 38
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 13 | 19 | 32
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 19 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 22 | 38

OUTCOME MEASURES:

1. Primary Outcome: Sympathetic Nerve Activity Burst Frequency
Description: Direct recordings of muscle sympathetic nerve activity (MSNA) from the peroneal nerve using a microelectrode.
Time Frame: 1 month
Population: 26 total participants were analyzed for primary outcome measures that completed both arms (fluid control vs. alcohol) of the study, using a randomized crossover design.
Measure: Mean (Standard Deviation); unit: Burst/Min
Groups:
- Fluid Control; Alcohol: All participants received both a binge alcohol dose (0.85g/kg for females, 1.0g/kg for males) and a fluid control drink (i.e., juice) of the same volume of fluid as the alcohol condition. These conditions were provided in a randomized, crossover design, and were separated by 1-month washout.
Arm/Group | Fluid Control | Alcohol
Number analyzed (Participants) | 26 | 26
Burst/Min | 18 (9) | 20 (8)
Statistical Analysis 1: Comparison: Fluid Control vs Alcohol; Statistical analysis on Burst Frequency (Burst/Min); Test type: Superiority — The original hypothesis was that resting MSNA burst frequency would be higher the morning after evening binge alcohol when compared to fluid control condition. A p-value of < 0.05 was used for significance; p = 0.283, t-test, 2 sided — The original hypothesis was that resting MSNA burst frequency would be higher the morning after evening binge alcohol when compared to fluid control condition. A p-value of < 0.05 was used for significance
Statistical Analysis 2: Comparison: Fluid Control vs Alcohol; Statistical analysis on Burst Incidence (Burst/100hb); Test type: Superiority — The original hypothesis was that resting MSNA burst incidence would be higher the morning after evening binge alcohol when compared to fluid control condition. A p-value of < 0.05 was used for significance; p = 0.920, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Sympathetic Nerve Activity Burst Incidence
Description: Direct recordings of muscle sympathetic nerve activity (MSNA) from the peroneal nerve using a microelectrode. Burst incidence is calculated as the number of sympathetic bursts per 100 heartbeats. This measure takes into account varying heart rates on sympathetic activity by normalizing to each individual's heartbeat. Higher calculated number equates to higher sympathetic activity.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: burst/100 heart beats
Arm/Group | Fluid Control | Alcohol
Number analyzed (Participants) | 26 | 26
burst/100 heart beats | 31 (16) | 31 (12)

3. Secondary Outcome: Spontaneous Sympathetic Baroreflex Sensitivity
Description: The linear relationship between beat-to-beat blood pressure and sympathetic nerve activity expressed as bursts/100 heart beats. Sympathetic baroreflex sensitivity is determined using the slope of the weighted linear regression of diastolic blood pressure and MSNA burst incidence. Diastolic blood pressure values of individual cardiac cycles were binned into 3 mmHg intervals, and the MSNA burst incidence was determined and subsequently plotted against corresponding diastolic blood pressure bins.
Time Frame: 1 month
Population: 11 total participants were analyzed for the secondary outcome measure that completed both arms of the study (fluid control vs. alcohol), with a randomized crossover design.
Measure: Mean (Standard Deviation); unit: MSNA Bursts/100 heart beats/mmHg
Arm/Group | Fluid Control | Alcohol
Number analyzed (Participants) | 11 | 11
MSNA Bursts/100 heart beats/mmHg | -2 (1) | -2 (1)
Statistical Analysis 1: Comparison: Fluid Control vs Alcohol; Test type: Superiority — The original hypothesis was that sympathetic baroreflex sensitivity would be blunted the morning after evening binge alcohol when compared to fluid control condition. A p-value of < 0.05 was used for significance; p = 0.888, t-test, 2 sided — The original hypothesis was that sympathetic baroreflex sensitivity would be blunted the morning after evening binge alcohol when compared to fluid control condition. A p-value of < 0.05 was used for significance

4. Other Pre Specified Outcome: Nocturnal Blood Pressure Dip
Description: Change in nocturnal blood pressure during sleep when compared to evening/morning wakefulness.
Time Frame: 1 month
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Sleep Quality
Description: Polysomnography will be used to determine the quality of sleep, with a primary focus on the apnea-hypopnea index.
Time Frame: 1 month
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Sympathetic Reactivity
Description: The change in muscle sympathetic nerve activity during an acute laboratory stressor.
Time Frame: 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: On average 1 to 2 months following initial laboratory testing session
Description: Participants were monitored for minor and serious adverse events throughout the protocol. Participants were not at risk for all-cause mortality and were not monitored for all-cause mortality. All participants were young healthy (male/female) adults and were screened for serious disorders that may predispose them towards unanticipated adverse events.
Arm/Group | Fluid Control | Alcohol
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 2/38 | 1/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluid Control (N=38) | Alcohol (N=38)
Nausea (Gastrointestinal disorders) | 0 | 1
Presyncope in response to venipuncture (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT03567434/Prot_SAP_ICF_000.pdf